CLINICAL TRIAL: NCT03239860
Title: A Long-Term International, Extension of Study GNC-003 With GNbAC1 in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Assessing the HERV-W Env ANtagonist GNbAC1 for Evaluation in an Open Label Long-term Safety Study in Patients With Multiple Sclerosis
Acronym: ANGEL-MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on R&D strategic reasons, our co-development Partner financing the study disengaged from the development of GNbAC1.
Sponsor: GeNeuro SA (Industry)
Collaborators: Les Laboratoires Servier (Unknown); Worldwide Clinical Trials (Other); Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-004
Record Dates: First submitted 2017-07-12; First posted 2017-08-04 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2018-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Multiple Sclerosis Relapsing-Remitting; GNbAC1; MRI; Monoclonal antibody; Multiple Sclerosis associated retrovirus MSRV; MS; RRMS; HERV-W; Temelimab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 GNbAC1 (Experimental): Monthly IV
  Interventions: Drug: GNbAC1 Monoclonal Antibody
- Dose 2 GNbAC1 (Experimental): Monthly IV
  Interventions: Drug: GNbAC1 Monoclonal Antibody
- Dose 3 GNbAC1 (Experimental): Monthly IV
  Interventions: Drug: GNbAC1 Monoclonal Antibody

INTERVENTIONS:
Drug: GNbAC1 Monoclonal Antibody — Monthly IV

SUMMARY:
The humanised IgG4 monoclonal antibody GNbAC1 targets the envelope protein (Env) of the human endogenous multiple sclerosis-associated retrovirus (HERV-W MSRV), which may play a critical role in multiple sclerosis.

The study assesses the long-term safety of GNbAC1 in patients with RRMS and the long-term efficacy of GNbAC1 in terms of MRI outcomes, relapse rate, disability and disease progression.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients must have completed Period 2 of study GNC-003 and must meet all eligibility criteria for the GNC-004 study
* Patients (male or female with reproductive potential) must agree to use highly effective methods of birth control
* Provision of written informed consent to participate prior to any trial procedure as shown by signature on the subject consent form.

Main Exclusion Criteria:

* Patients not having completed the study GNC-003
* Pregnancy
* The emergence of any disease diagnosis during the course of study GNC-003 that is not MS and could better explain the patient's neurological signs and symptoms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Long term safety of GNbAC1 | 96 Weeks
  The main parameters evaluated to assess the long term safety will be:
  AE and SAE, clinical safety laboratory, IgG4 dosing, vital signs, physical examination, ECGs, Anti-drug antibody and C-SSRS scale

SECONDARY OUTCOMES:
Long term efficacy of GNbAC1 in terms of MRI outcomes | 96 Weeks
Long term efficacy of GNbAC1 in terms of relapse rate | 96 Weeks
Long term efficacy of GNbAC1 in terms of disability | 96 Weeks
Long term efficacy of GNbAC1 in terms of disease progression | 96 Weeks

CONTACTS AND LOCATIONS:
Locations (12):
- Hospital, Sofia, Bulgaria
- Hospital, Zagreb, Croatia
- Hospital, Jihlava, Czechia
- Hospital, Tallinn, Estonia
- Hospital, Berlin, Germany
- Hospital, Budapest, Hungary
- Hospital, Rome, Italy
- Hospital, Warsaw, Poland
- Hospital, Moscow, Russia
- Hospital, Belgrade, Serbia
- Hospital, Barcelona, Spain
- Hospital, Kharkiv, Ukraine

REFERENCES:
- [Derived] Hartung HP, Derfuss T, Cree BA, Sormani MP, Selmaj K, Stutters J, Prados F, MacManus D, Schneble HM, Lambert E, Porchet H, Glanzman R, Warne D, Curtin F, Kornmann G, Buffet B, Kremer D, Kury P, Leppert D, Ruckle T, Barkhof F. Efficacy and safety of temelimab in multiple sclerosis: Results of a randomized phase 2b and extension study. Mult Scler. 2022 Mar;28(3):429-440. doi: 10.1177/13524585211024997. Epub 2021 Jul 9. PMID 34240656